CLINICAL TRIAL: NCT02211300
Title: MANUAL VS. AUTOMATED MONITORING ACCURACY OF GLUCOSE
Brief Title: MANAGE Automated Glucose Monitoring
Acronym: MANAGE IDE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: OptiScan Biomedical Corporation (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: Double | Purpose: Supportive Care
Other Study IDs: 2002055
Record Dates: First submitted 2014-06-17; First posted 2014-08-07 (Estimated); Last update posted 2015-06-29 (Estimated); Status verified 2015-06

CONDITIONS: ICU/CCU Patients Requiring Blood Glucose Monitoring
Keywords: glucose monitoring; OptiScanner

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Optiscanner values vs YSI (Experimental): Matched samples up to 12 times per 24 hour period
  Interventions: Device: The OptiScanner; Device: YSI 2300 STAT Plus™

INTERVENTIONS:
Device: The OptiScanner — treatment of blood glucose per standard of care
  Other Names: OptiScanner; Yellow Springs Instrument
Device: YSI 2300 STAT Plus™

SUMMARY:
The objective of this study is to demonstrate that the OptiScanner® is safe and can provide accurate blood glucose levels in critically ill subjects.

Accuracy Hypothesis:

The assessment of blood glucose level that results from the OptiScanner is comparable to the YSI 2300 STAT Plus™ Glucose and Lactate Analyzer ("YSI Analyzer"; YSI Life Sciences, Yellow Springs, OH).

Safety Hypothesis:

The OptiScanner has an acceptable risk/benefit profile for a system that can provide repeated automated blood glucose levels for critically ill subjects.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent by participant or his/her legally authorized representative
* At least 18 years old
* Admitted to the ICU or CCU
* Expected ICU or CCU stay of at least 18 hours at the time of enrollment (as judged by Investigator)
* Requires blood glucose monitoring; and
* A vascular access device that can be dedicated for connection to the OptiScanner is either already in-place, is planned to be placed for another purpose or can, in the opinion of the Investigator be safely placed exclusively for use in this study, and another access device is in place or can be placed for manually drawing samples to be evaluated using the YSI Analyzer. Note that CVCs should not be placed solely for the purposes of conducting this study. Refer to section 1.2.7 for details regarding vascular access devices and guidelines for selection and placement.

Exclusion Criteria:

* Pregnant or nursing
* In the Investigator's opinion the subject cannot safely tolerate the amount of saline required to be given to the subject (up to 360 mL per day)
* Hematocrit less than 15% or greater than 60%
* Subjects that require placement of an additional vascular access line will be excluded if they do not have a suitable access site free from any of the following conditions:

  * Peripheral vascular disease
  * History of placement site neuropathy or chronic pain
  * History of placement extremity coagulopathy or clot formation
  * History of vascular surgery on the same extremity as catheter placement
* Any medical condition that, in the Investigator's opinion, would warrant exclusion from the study or prevent the subject from completing the study, including but not limited to a high risk of complications associated with vascular access; or
* Participation in any other investigational drug or device study in the last 30 days and/or while enrolled in this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 230 (Estimated)
Dates: Start 2014-04; Primary Completion 2015-09 (Estimated); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
Primary Accuracy Endpoint | Accurancy up to 72 hours of monitoring per subject
  The mean absolute relative difference (MARD) in glucose level between the OptiScanner and the YSI Analyzer (average of 2 measures). To demonstrate accuracy the MARD must be less than or equal to 10%.

SECONDARY OUTCOMES:
Secondary Accuracy Endpoint | Accuracy up to 72 hours of subject monitoring
  The "population CV" will be computed as the standard deviation of the difference between the glucose level reported by the OptiScanner and the glucose level reported by the YSI Analyzer divided by the mean of the YSI Analyzer values. Repeated measures analyses will be used to account for possible correlation of measurements within patients. The population CV therefore gives an estimate of the extent of the effect of outliers on the accuracy estimation. If the "population CV" is less than 13%, the outcome of the secondary accuracy analysis will be considered a success.

OTHER OUTCOMES:
Number of Adverse events | up to 72 hours of subject monitoring

CONTACTS AND LOCATIONS:
Overall Officials: Grant V Bochicchio, MD, MPH, Principal Investigator — Washington University School of Medicine; Stanley A Nasraway, MD, Principal Investigator — Tufts Medical Center; Anthony Furnary, MD, Principal Investigator — Providence St. Vincents Medical Center; Linda Moore, MD, Principal Investigator — Hermann Memorial Hospital
Locations (4):
- United States (4):
  - Tufts Medical Center, Boston, Massachusetts
  - Washington University School of Medicine, St Louis, Missouri
  - Providence Heart and Vascular Institute, Portland, Oregon
  - Hermann Memorial Hospital, Houston, Texas

REFERENCES:
- [Derived] Nohra E, Buckman S, Bochicchio K, Chamieh J, Reese S, Merrill C, Schuerer D, Bochicchio GV. Results of a near continuous glucose monitoring technology in surgical intensive care and trauma. Contemp Clin Trials. 2016 Sep;50:1-4. doi: 10.1016/j.cct.2016.07.007. Epub 2016 Jul 6. PMID 27394384